CLINICAL TRIAL: NCT01541813
Title: Clinical, Biological, Genetic and Functional Characterization of Rare Iron Overload Phenotypes Associated With Hepcidin Deficiency Except C282Y Homozygosity.
Brief Title: Rare Iron Overloads Except C282Y Homozygosity : Description and Characterization.
Acronym: HEPCIDEF
Status: Terminated | Type: Observational
Why Stopped: rare overload and low recruitment
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Afssaps 201O-A00866-33
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-08

CONDITIONS: Rare Iron Overloads Except C282Y Homozygosity
Keywords: Rare iron overload; hepcidin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- iron overloads except C282Y homozygosity: Patients with an iron overloads except C282Y homozygosity

SUMMARY:
Chronic iron overload is responsible for morbidity and mortality. There are many genetic and acquired causes. One of them is an hepcidin deficiency. Hepcidin is the regulating hormone for iron. The study explores this specific cause, and aim to characterize this iron overload in term of clinical, biological, genetic and functional specificities.

DETAILED DESCRIPTION:
One of chronic iron overload profiles is a deficit in hepcidin. Hepcidin is the regulating hormone for iron. This specific profile is characterized by an elevated serum iron, an elevated transferrin saturation, and parenchymal damages of iron overload. This disease is not connected with known mutations of iron metabolism genes.

The main objective of this study is the clinical, biological, genetic and functional characterization of rare iron overload phenotypes associated with hepcidin deficiency except C282Y homozygosity.

ELIGIBILITY:
Inclusion criteria:

* Biological profile suggesting hepcidin deficiency:

  * high serum iron (> 25μmol / l) checked at least 2 times.
  * increased transferrin saturation coefficient (> 50 %) checked at least 2 times, and calculated from transferrinemia.
* Proved hepatic iron overload: using a dosage of iron hepatic concentration either on hepatic biopsy, or by MRI according to the method of iron overload quantification. A threshold of 100 µmol / g is set.
* Patient's written consent for examination and collection of genetic data to set the diagnosis.

Non inclusion criteria:

* HFE hemochromatosis: C282Y/C282Y homozygosity
* Treatment by iterative phlebotomies (more than 2 phlebotomies)
* Hematological diseases with dyserythropoiesis and/or repeated transfusions
* Low haptoglobin level, suggesting chronic hemolysis or myelodysplasia
* Long-term iron oral and/or parenteral supplementation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a rare iron overloads except C282Y homozygosity.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Bardou-Jacquet, MD, Principal Investigator — CHU Rennes
Locations (10):
- France (10):
  - Kremlin-Bicêtre Hospital, Le Kremlin-Bicêtre
  - CHRU - Huriez Hospital, Lille
  - Limoges CHU, Limoges
  - Lyon Sud Hospital, Lyon
  - Hospital of conception, Marseille
  - Saint Eloi Hospital - CHU, Montpellier
  - Emilie Muller Hospital, Mulhouse
  - Hospital Center, Mulhouse
  - BP 86709, Orléans
  - Purpan CHU, Toulouse